CLINICAL TRIAL: NCT02823249
Title: Effect of Amino Acids and Sugar Alcohols on Release of Satiation Peptides and Activation of Specific Brain Regions in Normal Weight and Obese Subjects
Brief Title: Effect of Amino Acids and Sugar Alcohols on Satiation Peptides and Activation of Specific Brain Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: fMRI Aminoacids
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases | interventions — Tryptophan; Leucine; Xylitol; Erythritol; Glucose; Proteins; CD36 Antigens; Carbohydrates; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1.56 g L-Tryptophan (Active Comparator): 1.56 g L-Tryptophan in 300 mL tap water given via nasogastric tube
  + after 60 min: 500ml of a mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate) given via nasogastric tube
  Interventions: Dietary Supplement: 1.56 g L-Tryptophan; Dietary Supplement: Tap water; Dietary Supplement: Mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate); Device: Nasogastric Tube
- 1.56 g L-Leucine (Active Comparator): 1.56 g L-Leucine in 300 mL tap water given via nasogastric tube
  + after 60 min: 500ml of a mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate) given via nasogastric tube
  Interventions: Dietary Supplement: 1.56 g L-Leucine; Dietary Supplement: Tap water; Dietary Supplement: Mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate); Device: Nasogastric Tube
- 50 g Xylitol (Active Comparator): 50 g Xylitol in 300 mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 50 g Xylitol; Dietary Supplement: Tap water; Device: Nasogastric Tube
- 75 g Erythritol (Active Comparator): 75 g Erythritol in 300 mL tap water given via nasogastric tube
  Interventions: Dietary Supplement: 75 g Erythritol; Dietary Supplement: Tap water; Device: Nasogastric Tube
- 75 g Glucose and mixed liquid meal (Placebo Comparator): 75 g Glucose in 300 mL tap water given via nasogastric tube
  + after 60 min: 500ml of a mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate) given via nasogastric tube
  Interventions: Dietary Supplement: 75 g Glucose; Dietary Supplement: Tap water; Dietary Supplement: Mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate); Device: Nasogastric Tube
- Tap water and mixed liquid meal (Placebo Comparator): 300 mL tap water given via nasogastric tube
  + after 60 min: 500ml of a mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate) given via nasogastric tube
  Interventions: Dietary Supplement: Tap water; Dietary Supplement: Mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate); Device: Nasogastric Tube

INTERVENTIONS:
Dietary Supplement: 1.56 g L-Tryptophan
  Arms: 1.56 g L-Tryptophan
Dietary Supplement: 1.56 g L-Leucine
  Arms: 1.56 g L-Leucine
Dietary Supplement: 50 g Xylitol
  Arms: 50 g Xylitol
Dietary Supplement: 75 g Erythritol
  Arms: 75 g Erythritol
Dietary Supplement: 75 g Glucose
  Arms: 75 g Glucose and mixed liquid meal
Dietary Supplement: Tap water
Dietary Supplement: Mixed liquid meal (Ensure Plus®; 17% protein, 29% fat and 54% carbohydrate)
  Arms: 1.56 g L-Leucine; 1.56 g L-Tryptophan; 75 g Glucose and mixed liquid meal; Tap water and mixed liquid meal
Device: Nasogastric Tube

SUMMARY:
With this study the investigators investigate the effects of amino acids (tryptophan, leucin) and sugar alcohols (xylitol, erythritol) on satiety mechanisms and brain activation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal weight subjects with a body-mass index of 19.0-24.9
* Healthy obese subjects with a body-mass index of > 30
* Normal eating habits (no diets; no dietary changes; no special dietary habits such as vegetarian/vegan)
* Age 18-40 years
* Stable body weight for at least three months

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medications (except for oral contraceptives)
* Medical or psychiatric illness
* History of gastrointestinal disorders
* Food allergies
* Pregnancy, breast feeding
* Body piercings that cannot be removed
* History of claustrophobia
* Left-hander

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effect of aminoacids on cerebral blood flow measured by functional brain MRI | changes from baseline to one hour after treatment
Effect of sugar alcohols on cerebral blood flow measured by functional brain MRI | changes from baseline to one hour after treatment

SECONDARY OUTCOMES:
Measurement of Plasma Glucose concentrations | changes from baseline to three hours after treatment
Measurement of Plasma Insulin concentrations | changes from baseline to three hours after treatment
Measurement of Plasma cholecystokinin concentrations | changes from baseline to three hours after treatment
Measurement of Plasma Glucagon-like Peptide (GLP-1) concentrations | changes from baseline to three hours after treatment
Measurement of Plasma PYY concentrations | changes from baseline to three hours after treatment
Measurement of Plasma ghrelin concentrations | changes from baseline to three hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided